CLINICAL TRIAL: NCT00477776
Title: Metoclopramide to Improve Lactogenesis II in Diabetic Women: a Randomized Controlled Trial
Brief Title: Maxolon to Improve Breastmilk Supply in Diabetic Women: a Randomised Controlled Trial
Acronym: Maxalon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: The University of Western Australia (Other)
Responsible Party: Professor Chong Yap Seng, National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHG SIG 06022
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Breastfeeding
Keywords: Beginning of breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- a (Active Comparator): Mother with diet-controlled diabetes receive Metoclopramide 10 mg 3 times a day for the first 7 days, and 2 times a day for day 8 to 10, and once a day from day 11 to day 12
  Interventions: Drug: Metoclopramide (Maxolon)
- b (Placebo Comparator): Placebo 10 mg 3 times a day for 7 days, 2 times a day from day 8 to day 10, and once a day for day 11 to 12
  Interventions: Drug: Placebo
- c (Active Comparator): Metoclopramide 10 mg 3 times a day for 7 days, 2 times a day from day 8 to day 10, and once a day from day 11 to 12
  Interventions: Drug: Metoclopramide (Maxolon)
- d (Placebo Comparator): Placebo 10 mg 3 times a day for 7 days, 2 times a day for day 8 to 10; and once a day from day 11 to 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide (Maxolon) — Metoclopramide 10 mg 3 times a day for 7 days, 2 times a day from day 8 to day 10, once a day for day 11 and 12
  Other Names: Maxalon
  Arms: a; c
Drug: Placebo — Placebo 10 mg 3 times a day for 7 days, 2 times a day from day 8 to 10, once a day from day 11 to 12
  Arms: b; d

SUMMARY:
Early use of oral maxalon can hasten and improve the establishment of breastfeeding in diabetic mothers after preterm and term deliveries.

Maxolon promotes breastfeeding by working on the central nervous system which increases the milk producing hormone, prolactin which in turn helps to increase the milk supply for breastfeeding. Successful early breastfeeding establishment is important for continued breastfeeding.

DETAILED DESCRIPTION:
The study aims to determine the breastfeeding initiation and duration rate of a cohort of pregnant women with gestational diabetes(diet-controlled) and insulin dependent and pre-existing diabetes, assess the impact of a post natally administered galactogogue, metoclopramide on the milk volume production and timing of lactogenesis II in diabetic women on diet control and insulin and determine the prolactin response to lactation among diabetic women on diet control and insulin.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with pregestational or gestational diabetes under diet or insulin control

Exclusion Criteria:

* Patient who have epilepsy or on anti-seizure medications,
* Patients who have a history of significant depression or are on antidepressant drugs
* Patients who have pheochromocytoma or uncontrolled hypertension
* Patients who have intestinal bleeding or obstruction
* Patient with known allergy or prior reaction to metoclopramide
* Patient with HIV infection
* Current pregnancy complicated by fetal congenital anomalies and multiple fetuses

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
a.successful initiation of lactation as determined by lactogenesis II markers, maternal perception and timing c.timing of successful establishment of lactogenesis II | within the first two weeks postpartum

SECONDARY OUTCOMES:
amount of breastmilk determined by testweighing and expressed milk volumes, weight change on day 7 and breastfeeding status up to 6 months | within 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Chong Y S, MBBS,MRACOG, Principal Investigator — National University Hospital and National University of Singapore; Citra Mattar, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Cregan MD, De Mello TR, Kershaw D, McDougall K, Hartmann PE. Initiation of lactation in women after preterm delivery. Acta Obstet Gynecol Scand. 2002 Sep;81(9):870-7. doi: 10.1034/j.1600-0412.2002.810913.x. PMID 12225305
- [Background] Hartmann PE, Cregan MD, Mitoulas LR. Maternal modulation of specific and non-specific immune components of colostrum and mature milk. Adv Nutr Res. 2001;10:365-87. doi: 10.1007/978-1-4615-0661-4_18. No abstract available. PMID 11795051
- [Background] Hartmann P, Cregan M. Lactogenesis and the effects of insulin-dependent diabetes mellitus and prematurity. J Nutr. 2001 Nov;131(11):3016S-20S. doi: 10.1093/jn/131.11.3016S. PMID 11694639
- [Background] Hansen WF, McAndrew S, Harris K, Zimmerman MB. Metoclopramide effect on breastfeeding the preterm infant: a randomized trial. Obstet Gynecol. 2005 Feb;105(2):383-9. doi: 10.1097/01.AOG.0000151113.33698.a8. PMID 15684169
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208